CLINICAL TRIAL: NCT01515566
Title: Effects of Prophylactic Subcutaneous Fentanyl on Exercise-Induced Breakthrough Dyspnea in Cancer Patients: A Preliminary Double-Blind, Randomized Controlled Trial
Brief Title: Breakthrough Dyspnea Fentanyl Study in Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2011-1007
Record Dates: First submitted 2012-01-13; First posted 2012-01-24 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Advanced Cancers; Dyspnea
Keywords: Advanced Cancer; Dyspnea; Exercise-induced breakthrough dyspnea; Shortness of breath; Fentanyl; Sublimaze; Placebo; Normal saline; NS; Questionnaires; Surveys; Walk test
MeSH Terms: conditions — Dyspnea | interventions — Fentanyl; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fentanyl (Experimental): Fentanyl subcutaneously (SQ) dose equivalent to 15-25% of the morphine equivalent daily dose (MEDD) 15 minutes before walk test, and 6 minute walk test (6MWT) at baseline and 15 minutes after Fentanyl. Two (2) Questionnaires completed at baseline taking about 10 minutes to complete, and one completed after study visit taking about 5 minutes to complete.
  Interventions: Drug: Fentanyl; Other: Walking Tests; Behavioral: Questionnaires
- Placebo (Active Comparator): Normal saline 0.9% preservative free SQ 15 minutes before walk test, and 6 minute walk test at baseline and 15 minutes after Placebo. Two (2) Questionnaires completed at baseline taking about 10 minutes to complete, and one completed after study visit taking about 5 minutes to complete.
  Interventions: Other: Placebo; Other: Walking Tests; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Fentanyl — Fentanyl SQ dose equivalent to 15-25% of the morphine equivalent daily dose (MEDD) 15 minutes before 6 minute walk test.
  Other Names: Sublimaze
  Arms: Fentanyl
Other: Placebo — Normal saline 0.9% preservative free SQ 15 minutes before walk test.
  Arms: Placebo
Other: Walking Tests — 6 minute walk test at baseline and 15 minutes after Fentanyl or Placebo.
Behavioral: Questionnaires — Questionnaires completed at baseline (two) and after study visit (one) taking about 5 ot 10 minutes to complete.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn if fentanyl given under the skin can reduce shortness of breath in cancer patients. Researchers also want to learn if it can help to improve your physical function. In this study, fentanyl will be compared to a placebo.

Fentanyl is commonly used for treatment of cancer pain. It is believed to help patients with their shortness of breath as well.

A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to either receive fentanyl or placebo. You will have an equal chance of being assigned to either group.

Study Drug/Placebo Administration:

Before you receive the study drug/placebo, you will walk back and forth in an indoor corridor for up to 6 minutes. You may feel out of breath or become exhausted. You may slow down, stop, and rest at any time you need to.

After that, you will sit down and rest (for up to 1 hour). During this time, the study drug/placebo will be prepared.

You will then be given a study drug/placebo shot under the skin in your arms or legs. You will then wait for another 15 minutes and repeat the walking test.

Study Visit:

During your study visit, the study staff will collect information from your medical record about your age, sex, race, disease type, how well you are able to perform the normal activities of daily living, any drugs you are taking, and possible causes of shortness of breath.

You will also complete 2 walking tests. Before the walk tests, you will complete 2 questionnaires. One (1) of them asks about any breathing symptoms you may be having, and the other asks about any other symptoms you may be having. It should take about 10 minutes to complete these questionnaires.

Before and after each walk test, the study staff will record your heart rate, breathing rate, and the level of air breathed out using a measuring device that will be clipped onto your finger. The study staff will also ask you questions about how hard it is to catch your breath and your level of tiredness.

During each walk test, you will be asked about how hard it is to catch your breath. The distance you walked and how often and for how long you stopped will be recorded. Before and after the second walk test, the study staff will ask you about any side effects from the study drug/placebo that you may be having.

During the rest period between the 2 walk tests, you may be asked how hard it is to catch your breath several times.

At the end of the study visit, you will fill out 1 questionnaire that asks if you think the study drug/placebo is helping you, and how satisfied you are with the study. It should take about 5 minutes to complete the questionnaire.

Length of Study:

You will be on this study for up to 100 minutes.You will be taken off study if intolerable side effects occur during the study.

This is an investigational study. Fentanyl is FDA approved and commercially available for the treatment of pain. It's use to help with shortness of breath is investigational.

Up to 20 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cancer
2. Breakthrough dyspnea, defined in this study as dyspnea on exertion with an average intensity level >=3/10 on the numeric rating scale
3. Outpatient or inpatient at MD Anderson Cancer Center seen by the Supportive Care or Rehabilitation Service
4. Able to communicate in English or Spanish
5. Ambulatory and able to walk with or without walking aid
6. On strong opioids with morphine equivalent daily dose of 30-580 mg, with stable (i.e. +/- 30%) regular dose over the last 24 hours
7. Karnofsky performance status >=50%
8. Age 18 or older

Exclusion Criteria:

1. Dyspnea at rest >=7/10 at the time of enrollment
2. Supplemental oxygen requirement >6 L per minute
3. Delirium (i.e. Memorial delirium rating scale >13)
4. History of unstable angina or myocardial infarction 1 month prior to study enrollment
5. Resting heart rate >120 at the time of study enrollment
6. Systolic pressure >180 mmHg or diastolic pressure >100 mmHg at the time of study enrollment
7. History of active substance abuse within the past 12 months
8. History of allergy to fentanyl
9. Unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hui D, Xu A, Frisbee-Hume S, Chisholm G, Morgado M, Reddy S, Bruera E. Effects of prophylactic subcutaneous fentanyl on exercise-induced breakthrough dyspnea in cancer patients: a preliminary double-blind, randomized, controlled trial. J Pain Symptom Manage. 2014 Feb;47(2):209-17. doi: 10.1016/j.jpainsymman.2013.03.017. Epub 2013 Jul 3. PMID 23830530
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient participants from the Supportive Care Center at MD Anderson Cancer Center were recruited between July 10, 2012 and December 12, 2012.
Pre-assignment Details: Six participants of the 26 recruited were excluded from the trial before assignment to groups due to ineligibility.
Groups:
- Fentanyl: Fentanyl subcutaneous (SQ) dose equivalent to 15-25% of the morphine equivalent daily dose (MEDD) 15 minutes before walk test; 6 minute walk test (6MWT) at baseline and 15 minutes after Fentanyl. Questionnaires completed at baseline and after study visit.
- Placebo: Normal saline 0.9% preservative free SQ 15 minutes before walk test; 6 minute walk test (6MWT) at baseline and 15 minutes after Placebo. Questionnaires completed at baseline and after study visit.
Period: Overall Study
Arm/Group | Fentanyl | Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fentanyl: Fentanyl SQ dose equivalent to 15-25% of the morphine equivalent daily dose (MEDD) 15 minutes before walk test; 6 minute walk test (6MWT) at baseline and 15 minutes after Fentanyl or Placebo. Questionnaires completed at baseline and after study visit.
- Placebo: Normal saline 0.9% preservative free SQ 15 minutes before walk test; 6MWT at baseline and 15 minutes after Fentanyl or Placebo. Questionnaires completed at baseline and after study visit.
- Total: Total of all reporting groups
Arm/Group | Fentanyl | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Secondary Outcome: Effect of Fentanyl Versus Placebo for Exercise-Induced and Breakthrough Dyspnea
Description: Participants receive either Fentanyl subcutaneous (SQ) 15 minutes before walking test, or Placebo (SQ) 15 minutes before walking test. During the study, trained research staff perform study assessments and monitor participant carefully throughout the study period. Six-minute walk tests were carried out following guidelines from the American Thoracic Society. The intensity of dyspnea at 0, 1, 2, 3, 4, 5 and 6 minute of each walk test were assessed using a validated numeric rating scale (NRS) ranging from 0 ("no shortness of breath") to 10 ("worst possible shortness of breath") and every 5 minutes during the rest period.
Time Frame: Baseline to 100 minutes for study participation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fentanyl: Fentanyl SQ dose equivalent to 15-25% of MEDD 15 minutes before walk test; 6MWT at baseline and 15 minutes after Fentanyl.
- Placebo: Normal saline 0.9% preservative free SQ 15 minutes before walk test; 6MWT at baseline and 15 minutes after Placebo.
Arm/Group | Fentanyl | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale
  Dyspnea at 0 minutes (Baseline walk test) | 2 (1) [1.8 to .4] | 3 (3) [1.5 to .1]
  Dyspnea at 6 minutes (Baseline walk test) | 6 (1) [3.2 to .4] | 7 (3) [4 to .02]
  Dyspnea at 0 minutes (Second walk test) | 1 (1) [1.8 to .04] | 2 (2) [1.5 to .1]
  Dyspnea at 6 minutes (Second walk test) | 4 (1) [3.2 to .4] | 5 (3) [4 to .02]

2. Primary Outcome: Retention Rate
Description: Retention rate is defined as the percentage of subjects able to complete the study.
Time Frame: Baseline to study completion, up to 100 minutes.
Measure: Number; unit: percentage of participants
Arm/Group | Fentanyl | Placebo
Number analyzed (Participants) | 10 | 10
percentage of participants | 100 | 100

3. Secondary Outcome: Effect of Fentanyl on Walk Distance
Description: Ambulatory patients with breakthrough dyspnea performed a baseline 6 minute walk test (6MWT), and then received either subcutaneous fentanyl or placebo 15 minutes before a second 6MWT. The change in walk distance was documented between the first and second 6MWT.
Time Frame: Baseline 6 minute walk test (6MWT) to second 6MWT, up to 100 minutes for study participation.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Fentanyl | Placebo
Number analyzed (Participants) | 10 | 10
feet
  Walk Distance (Baseline Walk Test) | 397.7 (98.1) | 399 (86.4)
  Walk Distance (Second Walk Test) | 434.9 (95.4) | 417.9 (89.3)

ADVERSE EVENTS:
Time Frame: Adverse effect collection from baseline up to 100 minutes for study participation.
Groups:
- Fentanyl: Fentanyl SQ dose equivalent to 15-25% of the morphine equivalent daily dose (MEDD) 15 minutes before walk test. 6 minute walk test at baseline and 15 minutes after Fentanyl.
- Placebo: Normal saline 0.9% preservative free SQ 15 minutes before walk test. 6 minute walk test at baseline and 15 minutes after Placebo.
Arm/Group | Fentanyl | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fentanyl (N=10) | Placebo (N=10)
Pain with subcutaneous injection (General disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The small sample size means findings are susceptible to random errors and regression to the mean.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes